CLINICAL TRIAL: NCT06205667
Title: Computer Guided Versus Conventional Arthrocentesis in Management of Internal Derangements: A Randomized Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FD-ASU-RCC.IM022204
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2021-03

CONDITIONS: TMJ - Oral &Maxillofacial Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer Guided Arthrocentesis (Experimental): a study group injected intra-articularly through TMJ using a computer-guided template.
  Interventions: Procedure: Computer Guided Arthrocentesis
- Conventional Arthrocentesis (Active Comparator): a control group which injected intra-articular through TMJ using conventional method based on anatomical landmark determination
  Interventions: Procedure: Conventional Arthrocentesis

INTERVENTIONS:
Procedure: Computer Guided Arthrocentesis — patients are going to be injected intra-articular within the superior joint space of the affected TMJ through custom guided template planned in a manner inspired by earphone design to get support from the tragus.
  Arms: Computer Guided Arthrocentesis
Procedure: Conventional Arthrocentesis — patients are going to be injected intra-articular within the superior joint space of the affected TMJ using conventional method anatomical landmark determination
  Arms: Conventional Arthrocentesis

SUMMARY:
The aim of the study is to evaluate the applicability, accuracy, benefits and the efficacy of 3-dimensional, printed, patient-specific guides to direct TMJ access for arthrocentesis when performed in contrast with conventional arthrocentesis of TMJ.

ELIGIBILITY:
Inclusion Criteria:

* Patients who complain from signs and symptoms of internal derangements and were diagnosed by the RDC/TMD as having disc displacement with/ without reduction with / without limitation associated with arthralgia or as having disc displacement with reduction associated with arthralgia in a presence or absence of joint sounds.
* Patients who did not responded to conservative treatment for a minimum of 3 months.
* Obtaining written informed consents signed by the patients.

Exclusion Criteria:

* Patients suffering from any muscular disorders as myofascial pain or myofascial pain with limitations
* If the disc was not visible in the MRI examination.
* Patients who previously received intra-articular injection of any medication or exposed to any other TMJ invasive procedure.
* Patients who suffer from any connective tissue diseases as rheumatoid arthritis or neurologic disorders.
* Patients with history of major jaw trauma, bisphosphonate-derived drug use, pregnancy, alcohol or drug dependence.
* Patients with gross mechanical restrictions or history of adhesion (fibrous or bony).
* Patients with psychiatric disease or substance abuse or have an allergy to the substance used in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Attempts number of needle puncture | intraoperative
Operation time started from first needle insertion. | intaoperative

SECONDARY OUTCOMES:
Maximum mouth opening | 1week, 1, 3 and 6
  Change of mouth opening measurement using RDC/TMD
Pain reduction | 1week, 1, 3 and 6
  Pain assessment using Visual analogue Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams university, Cairo, Egypt